CLINICAL TRIAL: NCT03853265
Title: The Effect Of Virtual Reality Glasses On The Behavior Of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: HM20015131
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Study is parallel design with control group having the option of receiving treatment after study data is collected from initial treatment group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Virtual Reality (Experimental): Simulated dental office visit
  Interventions: Behavioral: Simulated dental office visit

INTERVENTIONS:
Behavioral: Simulated dental office visit — An immersive first-person point of view (POV) video simulation of the dental office in the three-dimensional environment (using a virtual reality headset) which allows participant to look around the room as they move down the hallways which is to be watched/experienced by the participant as often as possible between the initial visit and the follow up visit
  Arms: Virtual Reality

SUMMARY:
The aim of this study is to determine whether the use of virtual reality glasses showing an immersive video simulation of the dental visit will help decrease anxiety at future appointments by decreasing the element of surprise and increasing the patient's familiarity and comfort level with a specific dental practice environment.

DETAILED DESCRIPTION:
After an initial baseline data collection visit to the dental clinic, patients will be placed in the virtual reality (VR) group or the no VR group. Caregivers in the VR group will be given VR glasses. They will be instructed how to access the video and use the glasses. The child/wearer of the glasses will feel immersed in the three-dimensional environment and be able to look around the room as they move down the hallways in the video. The caregiver will be encouraged to have the child wear the VR glasses as often as possible and record the number of times the video is watched. The caregiver will fill out a "records form" which will include the date and time the video was watched. Both groups will then return to the clinic for follow up data collection visit.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder (ASD)

Exclusion Criteria:

* No specific diagnosis of Autism Spectrum Disorder (ASD)
* Limited English Proficiency
* Existing patient of VCU Department of Pediatric Dentistry
* Parent/guardian determination that child would not be avle to tolerate immersive simulation with VR glasses

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Change in heart rate | Baseline to 2 week follow up
  Heart rate measured by a fitbit worn on the wrist during the visit
Change in 5-point Venham Anxiety Scores | Baseline to 2 week follow up
  Level of Anxiety exhibited by participant during dental visit as rated on Venham Anxiety Scale by blinded expert rater. Scale ranges from 0 (relaxed, smiling, willing and able to converse) to 5 (child out of contact with the reality of the threat, loud crying, unable to listen to verbal communication, actively involved in escape behavior).
Change in 5-point Venham Uncooperative Behavior Scores | Baseline to 2 week follow up
  Cooperative behaviors exhibited by participant during dental visit as rated on Venham Uncooperative Behavior Scale by blinded expert rater. Scale ranges from 0 (total cooperation, no crying or physical protest) to 5 (general protest, no compliance or cooperation)

CONTACTS AND LOCATIONS:
Overall Officials: Tegwyn Brickhouse, DDS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No